CLINICAL TRIAL: NCT01720563
Title: A Phase II Double-blind and Randomized Trial Comparing Concurrent Chemoradiotherapy Plus PG2 Injection Versus Concurrent Chemoradiotherapy Plus Placebo in Advanced Pharyngeal or Laryngeal Squamous Cell Carcinoma
Brief Title: A Phase II Trial of PG2 in Patients With Advanced Pharyngeal or Laryngeal Squamous Cell Carcinoma Under Concurrent Chemoradiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change study drug dosage form
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PH-CP021
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Cancer-related Fatigue
Keywords: Cancer-related fatigue; astragalus polysaccharides; concurrent chemoradiotherapy; squamous cell carcinoma of head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Chemoradiotherapy; Cisplatin; Tegafur; Uracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Procedure: Concurrent chemoradiotherapy with PUL (cisplatin/tegafur plus uracil (UFT)/leucovorin) every 2 weeks
- Treatment (Experimental): Astragalus polysaccharides 500 mg
  Interventions: Drug: Astragalus polysaccharides 500 mg; Procedure: Concurrent chemoradiotherapy with PUL (cisplatin/tegafur plus uracil (UFT)/leucovorin) every 2 weeks

INTERVENTIONS:
Drug: Astragalus polysaccharides 500 mg — PG2 (500 mg in 500 ml saline), t.i.w. via i.v. infusion for 2.5-3.5 hours during the CCRT
  Other Names: PG2 Injection 500 mg
  Arms: Treatment
Drug: Placebo — 500 ml saline, t.i.w. via i.v. infusion for 2.5-3.5 hours during the CCRT
  Arms: Control
Procedure: Concurrent chemoradiotherapy with PUL (cisplatin/tegafur plus uracil (UFT)/leucovorin) every 2 weeks

SUMMARY:
Eighty to 90% of SCCHN (squamous cell carcinoma of head and neck) patients in Taiwan were betel quid chewers. Thirty to 40% of them experienced mucositis World Health Organization (WHO) grade 3 from cisplatin/flurouracil (FU) in neoadjuvant chemotherapy setting. This was higher than the 8-11% reported in the Western populations and was related to oral submucous fibrosis from betel quid chewing.Severer toxicities, esp. mucositis, could be anticipated in patients of betel quid chewing treated by concurrent chemoradiotherapy (CCRT) with cisplatin/FU.PG2 Injection is proved to be safe for clinical use and is effective in stimulating the recovery of hematopoiesis and immunity from chemotherapy-induced myelosuppression. It also improved the Quality of Life, especially in fatigue, among advanced cancer patients. This study will be investigated the effect of PG2 Injection in relieving the adverse events of concurrent chemoradiotherapy, such as fatigue, myelosuppression, mucositis, body weight loss, and even the compliance of radiotherapy and chemotherapy in treatment of patients with advanced pharyngeal or laryngeal SCCHN.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of squamous cell carcinoma
* Primary tumor site in the head and neck area
* Stage III or IV disease
* Measurable locoregional disease and no distant metastasis
* No prior cancer treatment
* 20-70 years old
* KPS ≧ 70
* Adequate bone marrow, liver, and renal function
* Fed with gastric tubes but without intestinal malabsorption or obstruction
* Not pregnancy and use a reliable contraceptive method during the study
* Signed informed consent
* Willing and able to complete quality of life questionnaires

Exclusion Criteria:

* Decompensated liver function
* Serious concomitant illness that might be aggravated by chemotherapy
* Active cardiac disease preceding the entry into the study
* Severe uncontrolled hypertension
* Uncontrolled infection
* History of other malignancy
* Pregnant or breast feeding
* Receiving other concomitant chemotherapy, radiotherapy or any other anticancer treatment
* Mental status not suitable for clinical trials
* Intestinal obstruction or malabsorption.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Fatigue status by Brief Fatigue Inventory (BFI) | 8 weeks

SECONDARY OUTCOMES:
Symptoms/Quality of Life Assessments by EORTC (European Organisation for Research and Treatment of Cancer) QLQ-C30 and H&N 35 questionnaires | 8 weeks
Karnofsky Performance Scale (KPS) | 8 weeks
Incidences of myelosuppression | 8 weeks
Serum inflammatory cytokines and c-reactive protein | 8 weeks
Weight loss | 8 weeks
Incidence of adverse events | 8 weeks
Tumor response | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Ming HM Wang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan